CLINICAL TRIAL: NCT02306291
Title: A Phase I/II, Open-label Multicenter Trial to Determine Safety, Pharmacokinetics and Efficacy of GMI-1271 in Combination With Chemotherapy in Patients With Acute Myeloid Leukemia
Brief Title: Study to Determine Safety, Pharmacokinetics and Efficacy of GMI-1271 in Combination With Chemotherapy in AML
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GMI-1271-201
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: AML; Acute myeloid leukemia; E-selectin; relapse refractory; elderly newly diagnosed; induction
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — uproleselan; Mitoxantrone; Etoposide; Cytarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Phase I) (Experimental): GMI-1271 in combination with mitoxantrone, etoposide and cytarabine (MEC) in relapsed/refractory subjects 18 years and older
  Interventions: Drug: GMI-1271; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine
- Arm B (Phase II Arm A) (Experimental): GMI-1271 in combination with mitoxantrone, etoposide and cytarabine (MEC) in relapsed/refractory subjects 18 years and older
  Interventions: Drug: GMI-1271; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine
- Arm C (Phase II Arm B) (Experimental): GMI-1271 in combination with cytarabine and idarubicin (7+3 regimen) in newly diagnosed subjects 60 years and older
  Interventions: Drug: GMI-1271; Drug: Cytarabine; Drug: Idarubicin

INTERVENTIONS:
Drug: GMI-1271 — E-selectin antagonist
  Other Names: Uproleselan
Drug: Mitoxantrone — induction chemotherapy
  Arms: Arm A (Phase I); Arm B (Phase II Arm A)
Drug: Etoposide — induction chemotherapy
  Arms: Arm A (Phase I); Arm B (Phase II Arm A)
Drug: Cytarabine — induction chemotherapy
Drug: Idarubicin — induction chemotherapy
  Arms: Arm C (Phase II Arm B)

SUMMARY:
This study will evaluate GMI-1271, a specific E-selectin antagonist, in acute myeloid leukemia in combination with standard agents used to treat this disease.

ELIGIBILITY:
Inclusion criteria:

1. AML (including secondary AML) diagnosed as per WHO criteria
2. For relapsed/refractory subjects only:

   * Subjects age ≥ 18 years with relapsed or refractory AML after ≤ 2 prior induction regimens, at least one containing anthracyclines
   * Medically eligible to receive MEC
   * Absolute blast count (ABC) ≤ 40,000/mm
3. For treatment-naïve subjects only:

   * Subjects ≥ 60 years of age with newly diagnosed AML
   * Medically eligible to receive "7+3" cytarabine/idarubicin
   * ABC count ≤ 40,000/mm
4. ECOG performance status 0-2
5. Hemodynamically stable and adequate organ function

Exclusion criteria:

1. Acute promyelocytic leukemia
2. Acute leukemia of ambiguous lineage (biphenotypic leukemia)
3. Active signs or symptoms of CNS involvement by malignancy
4. No prior G-CSF, GM-CSF or plerixafor within 14 days of study drug dosing
5. Known history or evidence of active hepatitis A, B, or C or HIV
6. Uncontrolled acute life threatening bacterial, viral or fungal infection
7. Active graft versus host disease (GVHD) ≥ Grade 2 or extensive chronic GVHD requiring immunosuppressive therapy
8. Hematopoietic stem cell transplantation ≤ 4 months of dosing
9. Clinically significant cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Safety assessed by frequency, severity and relatedness of adverse events | up to 44 days

SECONDARY OUTCOMES:
Time versus plasma concentration profile of GMI-1271 | up to 11 days
  Plasma concentration of GMI-1271
Overall response rate | up to 12 months
  Proportion of subjects who achieve a complete response (CR) or CR with incomplete blood count recovery (CRi) per local investigator assessment
Time to response | up to 12 months
  Time from date of first dose to first documentation of response
Duration of response | up to 12 months
  Time from date of first documented remission to the date of relapse or death from any cause, whichever occurs first
Event-free survival | up to 12 months
  Time from date of first dose to the date of treatment failure, relapse, or death from any cause, whichever occurs first
Overall survival | up to 12 months
  The probability of survival at 6 months (Phase 1) and 12 months (Phase 2), after the date of first dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Daniel DeAngelo, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (6):
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Ann Arbor, Michigan
  - University of Rochester, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Washington, Seattle, Washington
- Princess Alexandra Hospital, Brisbane, Australia
- University Hospital Galway, Galway, Ireland

REFERENCES:
- [Derived] DeAngelo DJ, Jonas BA, Liesveld JL, Bixby DL, Advani AS, Marlton P, Magnani JL, Thackray HM, Feldman EJ, O'Dwyer ME, Becker PS. Phase 1/2 study of uproleselan added to chemotherapy in patients with relapsed or refractory acute myeloid leukemia. Blood. 2022 Feb 24;139(8):1135-1146. doi: 10.1182/blood.2021010721. PMID 34543383